CLINICAL TRIAL: NCT00919568
Title: Arrhythmia Detection With Adherent Patient Monitoring
Brief Title: Monitoring Arrhythmia Patients (IMPACT)
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat, VP Clinical and Regulatory affairs, Corventis
Other Study IDs: COR-2009-005
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, multicenter, non-randomized study to determine the performance of NUVANT Mobile Cardiac Telemetry system in arrhythmia detection.

DETAILED DESCRIPTION:
Arrhythmia patients will be externally monitored. The collected information will be used to evaluate the NUVANT MCT system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing remote ambulatory electrocardiographic monitoring

Exclusion Criteria:

* Is participating in another clinical study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Remote cardiac monitoring
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Corventis, Inc.
Locations (1):
- Dr. Bedi, Steubenville, Ohio, United States